CLINICAL TRIAL: NCT04249232
Title: Abaloparatide Versus Placebo for Pelvic Fracture Healing - A Phase 2 Randomized Controlled Trial
Brief Title: Abaloparatide and Pelvic Fracture Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Weill Medical College of Cornell University (Other); Icahn School of Medicine at Mount Sinai (Other); New York University (Other); Westchester Medical Center (Other)
Responsible Party: Principal Investigator, Jeri Nieves, PhD, Professor of Clinical Epidemiology and Senior Research Scientist, Hospital for Special Surgery, New York
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-1978
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Fracture of Pelvis (Disorder)
Keywords: abaloparatide
MeSH Terms: conditions — Hip Fractures | interventions — abaloparatide

STUDY DESIGN:
Intervention Model Description: Parallel assignment with randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- abaloparatide prefilled syringe (Active Comparator): Abaloparatide-SC is supplied as a liquid, 3120 micrograms per 1.56 milliliter (2000 mcg/mL) in a single patient multi-use prefilled pen. The prefilled pen delivers 30 doses of abaloparatide, each containing 80 mcg of abaloparatide in 40 microliters of a sterile, clear, colorless solution. To be administered subcutaneously daily.
  Interventions: Drug: Abaloparatide 80 micrograms per Pen dose
- Placebo prefilled syringe (Placebo Comparator): For the placebo-SC a prefilled multi-use pen injector cartridge is designed to deliver 30 doses of placebo each in 40 microliters of sterile, clear, colorless solution to be administered subcutaneously daily.
  Interventions: Drug: Placebo prefilled injector pen

INTERVENTIONS:
Drug: Abaloparatide 80 micrograms per Pen dose — prefilled injector pen to deliver 80 micrograms daily subcutaneously
  Other Names: Tymlos
  Arms: abaloparatide prefilled syringe
Drug: Placebo prefilled injector pen — prefilled injector pen to deliver inactive solution daily subcutaneously
  Other Names: placebo
  Arms: Placebo prefilled syringe

SUMMARY:
This is a prospective randomized, double-blinded, placebo-controlled, phase 2, three-month study of the efficacy of abaloparatide in postmenopausal women and men ≥ 50 years of age with acute fractures of the pelvis (n=78). The primary outcome is CT image based evidence of fracture healing. The secondary aims are pain and physical performance measures at 3 months. This study will be extended with 9 months of open label abaloparatide to determine if any potential differences between the placebo and abaloparatide groups during the 3 months of treatment are evident and persist over time, even in patients who use abaloparatide after the three-month placebo controlled intervention.

DETAILED DESCRIPTION:
By 2030 over 25% of the entire US population will be older than 65 years of age. Pelvic fracture rates are higher in women. Over 90% of pelvic fractures in patients >60 years are defined as osteoporosis related fractures. In a recent study in Germany, the rate of all first pelvic fractures in persons over 60 was 22.4 [95% CI 22.0-22.9] per 10,000 person-years. The incidence rate increases dramatically with age, from 5.4 and 3.8 per 10,000 person-years in women and men aged 65 to 69 years to 93.5 and 44.5 per 10,000 person-years in women and men aged 90 years and older, respectively. This is in agreement with studies in the US and Finland, also showing an increase in incidence of pelvic fractures with age. Pelvic fractures are most often a result of low-energy trauma, such as a fall from standing height. Pelvic fractures are the most relevant for this proposed randomized placebo-controlled study. This fracture is accompanied by severe pain, chronic immobility and loss of function and independence in the elderly. The current treatment strategy of pelvic fractures includes pain management, patient mobilization, and the prevention of complications associated with comorbid conditions. In a review of six studies with over 500 patients, the mean length of hospital stay was 13.4 days and the average 1-year mortality was 16.3%. Mortality rates in 1300 pelvic fracture patients were still elevated at 3 years. Pelvic fractures are associated with slow healing and a delayed return to full function and normal activity. Pelvic fractures consume substantial healthcare resources, and based on administrative claims data, they are one of the most costly osteoporosis related fractures. Un-healed fractures, occurring in one-third of pelvic fracture patients at 3 months, can cause continued pain and impact mobility. With aging of the population and expected concomitant increase in the incidence of pelvic fractures, there is a pressing need to find effective treatments that will accelerate healing. There are strong preclinical data, as well as clinical evidence, that administration of parathyroid hormone (PTH) receptor agonists may improve bone union, hasten fracture healing and improve physical function. In one nonrandomized, un-blinded study, 100% of pelvic fracture patients given 1-84PTH were healed within 12 weeks compared to 68% of the controls. However, there is not sufficient evidence at this time to recommend routine use of PTH receptor agonists for fracture healing. Pelvic fractures are ideal to study for the impact of abaloparatide on rate of fracture healing because there are no surgical repairs for the vast majority of the fractures. Prior studies of teriparatide on wrist fracture healing were limited and confounded by the increased prevalence of surgical fixation to treat these fractures. Strong evidence of pelvic fracture healing that may result from this study may not only have an impact on pelvic fractures but perhaps may indicate a potential use for other fractures as well.

In the proposed randomized, double blind, placebo controlled clinical trial in patients >50 years of age with acute pelvic fracture, the investigators plan to evaluate whether treatment with daily subcutaneous ABALOPARATIDE 80 mcg/day compared with placebo, in addition to standard treatment (pain management, bed rest and prevention of complications from comorbid conditions), is effective in accelerating fracture healing in women and men compared to standard treatment alone. The investigators hypothesize that development of a successful adjunctive therapy (ABALOPARATIDE) will accelerate radiographic evidence of fracture healing and speed functional recovery. If this hypothesis holds true, it would lead to a change in clinical practice and an improved quality of care for pelvic fracture patients. Evidence of an impact on the healing of pelvic fractures may also extend to a potential to improve healing of other osteoporosis-related fractures. In the planned trial the investigators will recruit women and men with acute pelvic fractures and address 3 specific aims over 3 months of treatment in a placebo controlled double blind study to determine if ABALOPARATIDE in addition to standard care versus placebo and standard care:

1. Results in evidence of more complete cortical bridging at 3 months using focus CT to reduce radiation exposure from CT scans (primary outcome).
2. Leads to a faster reduction in pain as assessed by both the Numeric Rating Scale and a reduction in the use of narcotics (secondary outcome).
3. Leads more to a more rapidly improved functional outcome using measures to assess lower extremity function (Continuous Summary Physical Performance Score and Timed Up and Go- secondary outcomes).

Although the primary analysis will be based on data from 0 to 3 months, whether the benefit of ABALOPARATIDE on fracture healing wanes over time is unclear, making a longer follow-up important to extend knowledge on the persistence of early ABALOPARATIDE effect on these outcomes. Therefore, the investigators will extend this study with 9 months of open label ABALOPARATIDE to determine if any potential differences between the placebo and ABALOPARATIDE groups during the 3 months of treatment are evident and persist over time, even in patients who use ABALOPARATIDE after the three month placebo controlled intervention.

If ABALOPARATIDE can improve fracture healing, this study will have an impact on the treatment of persons with pelvic fracture who are not surgical candidates and often face severe pain, chronic immobility, and loss of function in the elderly. A positive finding of accelerated healing of pelvic fractures would also encourage study of ABALOPARATIDE for treatment of other osteoporotic fractures.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women and men >50 years of age with acute pelvic fractures, occurring with minimal trauma, presenting to Mount Sinai, New York University, New York Presbyterian-Queens, Hospital for Special Surgery, or New York Hospital (Cornell Medical) within one month of the onset of symptoms.

Exclusion Criteria:

1. Persons unable to complete the NRS and other surveys based on assessment by the study doctor.
2. Previously (prior to fracture) non-ambulatory subjects
3. Exclusion criteria related to contraindication or intolerance to ABALOPARATIDE:

   1. Hypersensitivity to ABALOPARATIDE
   2. Patients with increased risk of osteosarcoma: Paget's disease, history of radiation treatment
   3. Patients with active hypercalcemia based on serum calcium above the upper limit of normal.
   4. Serum creatinine cannot be elevated more than 1.5 times above upper normal limit for age
   5. Current diagnosis of hyperparathyroidism and other metabolic bone disease including osteogenesis imperfecta
   6. Multiple Kidney stones (calcium oxalate) within the last 10 years or single kidney stone (calcium oxalate) within the last year. If stone type is not known, a 24-hour urine calcium determination can be performed; if not elevated, the patient does not require exclusion.
   7. Normal alkaline phosphatase levels will not be used as an entrance criterion because most fracture patients will have elevations due to the acute fracture. However, we will attempt to obtain lab tests from the period prior to fracture to determine if they were normal. If unexplained elevations in alkaline phosphatase (more than 1.5 times above the upper limit of normal) are found in labs prior to the fracture, we will exclude that subject.
   8. Diagnosis of metastatic cancer within the past 10 years; primary bone cancer or multiple myeloma at any time. For other primary active non-skin cancers (diagnosed within the last 5 years), the patient's oncologist should be consulted to determine participant eligibility.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Efficacy for fracture healing- Measured by participant cortical bridging scores | 3 months
  Score for cortical bridging on a CT exam at 3 months in abaloparatide versus placebo groups.

SECONDARY OUTCOMES:
Efficacy measure of participant pain score as assessed by the Numeric Rating Scale | 8 weeks
  Pain score measured by Numeric rating scale that uses a scale from 0 (no pain) to 10 (worst pain imaginable), the subject will report how intense their pain is now and how intense it was on average last week. This will be compared in the abaloparatide versus placebo groups.
Efficacy measure of participant pain score as assessed by the Numeric Rating Scale | 12 months
  Pain score measured by Numeric rating scale that uses a scale from 0 (no pain) to 10 (worst pain imaginable), the subject will report how intense their pain is now and how intense it was on average last week. This will be compared over time in the abaloparatide versus placebo groups.
Participant lower extremity function based on a score from the Continuous Summary Physical Performance Score. The measure of lower extremity physical function is an efficacy variable. | 3 months
  Physical function as an efficacy outcome using a continuous summary physical performance score based on a battery of tests, including walk speed, repeated chair stands and balance.
Participant lower extremity function based on a score from the Continuous Summary Physical Performance Score. The measure of lower extremity physical function is an efficacy variable. | 12 months
  Physical function as an efficacy outcome using a continuous summary physical performance score based on a battery of tests, including walk speed, repeated chair stands and balance.
Participant (percent) reporting narcotic use for pain | 8 weeks
  The use of narcotics will be collected at each visit and will be quantified into morphine equivalents. ABALOPARATIDE versus placebo groups will be compared for morphine equivalents.
Efficacy measure of the time for participants to complete the Timed Up and Go Test. | 3 months
  The test begins by having the subject Stand up from the chair, walk to the line on the floor at a normal pace, turn, walk back to the chair at a normal pace and sit down again. The person administering the test will time the subject using a stopwatch.
  including walk speed, repeated chair stands and balance. In addition,Timed up and go score.

CONTACTS AND LOCATIONS:
Overall Officials: Jeri W Nieves, PhD, Principal Investigator — Hospital for Special Surgery, New York; Joseph Lane, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (3):
- United States (3):
  - Hospital for Special Surgery, New York, New York
  - Mount Sinai, New York, New York
  - Westchester Medical Center, Valhalla, New York

IPD SHARING:
Plan to Share IPD: Yes
Research data is identified by an anonymous study identification. No protected health information is stored in the research database. The possibility of individual subject identification is nil from within the purview of the data. The data will be made available for sharing 12-months after the publication of the primary paper. SAS datasets, a data dictionary, images of case report forms, SAS format library, the SAS program in which source data is recoded for analysis and data table summary descriptive statistics for data validation cross-check will be made available on an encrypted USB drive. A data sharing agreement is required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within one year of study completion
Access Criteria: A data sharing agreement is required. Dr. Nieves and Dr. Lane will give priority to data sharing requests with the stated purpose of a) Teaching, b) replication or reanalysis of results reported in the primary paper, c) subgroup analyses to be used for the design of future research. Other requests will be considered on a caseby- case basis. Hospital for Special Surgery legal office for research will provide details on their policy.

REFERENCES:
- [Background] Prieto-Alhambra D, Aviles FF, Judge A, Van Staa T, Nogues X, Arden NK, Diez-Perez A, Cooper C, Javaid MK. Burden of pelvis fracture: a population-based study of incidence, hospitalisation and mortality. Osteoporos Int. 2012 Dec;23(12):2797-803. doi: 10.1007/s00198-012-1907-z. Epub 2012 Feb 4. PMID 22310957
- [Background] Kannus P, Palvanen M, Niemi S, Parkkari J, Jarvinen M. Epidemiology of osteoporotic pelvic fractures in elderly people in Finland: sharp increase in 1970-1997 and alarming projections for the new millennium. Osteoporos Int. 2000;11(5):443-8. doi: 10.1007/s001980070112. PMID 10912847
- [Background] Andrich S, Haastert B, Neuhaus E, Neidert K, Arend W, Ohmann C, Grebe J, Vogt A, Jungbluth P, Rosler G, Windolf J, Icks A. Epidemiology of Pelvic Fractures in Germany: Considerably High Incidence Rates among Older People. PLoS One. 2015 Sep 29;10(9):e0139078. doi: 10.1371/journal.pone.0139078. eCollection 2015. PMID 26418971
- [Background] Benzinger P, Becker C, Kerse N, Bleibler F, Buchele G, Icks A, Rapp K. Pelvic fracture rates in community-living people with and without disability and in residents of nursing homes. J Am Med Dir Assoc. 2013 Sep;14(9):673-8. doi: 10.1016/j.jamda.2013.03.012. Epub 2013 May 13. PMID 23680402
- [Background] Melton LJ 3rd, Sampson JM, Morrey BF, Ilstrup DM. Epidemiologic features of pelvic fractures. Clin Orthop Relat Res. 1981 Mar-Apr;(155):43-7. PMID 7226629
- [Background] Alnaib M, Waters S, Shanshal Y, Caplan N, Jones S, St Clair Gibson A, Kader D. Combined pubic rami and sacral osteoporotic fractures: a prospective study. J Orthop Traumatol. 2012 Jun;13(2):97-103. doi: 10.1007/s10195-012-0182-2. Epub 2012 Mar 6. PMID 22391943
- [Background] Krappinger D, Kammerlander C, Hak DJ, Blauth M. Low-energy osteoporotic pelvic fractures. Arch Orthop Trauma Surg. 2010 Sep;130(9):1167-75. doi: 10.1007/s00402-010-1108-1. Epub 2010 Jun 3. PMID 20521061
- [Background] Peichl P, Holzer LA, Maier R, Holzer G. Parathyroid hormone 1-84 accelerates fracture-healing in pubic bones of elderly osteoporotic women. J Bone Joint Surg Am. 2011 Sep 7;93(17):1583-7. doi: 10.2106/JBJS.J.01379. PMID 21915572
- [Background] Ellegaard M, Jorgensen NR, Schwarz P. Parathyroid hormone and bone healing. Calcif Tissue Int. 2010 Jul;87(1):1-13. doi: 10.1007/s00223-010-9360-5. Epub 2010 Apr 29. PMID 20428858
- [Background] Goldhahn J, Feron JM, Kanis J, Papapoulos S, Reginster JY, Rizzoli R, Dere W, Mitlak B, Tsouderos Y, Boonen S. Implications for fracture healing of current and new osteoporosis treatments: an ESCEO consensus paper. Calcif Tissue Int. 2012 May;90(5):343-53. doi: 10.1007/s00223-012-9587-4. Epub 2012 Mar 28. PMID 22451221
- [Background] Aspenberg P, Genant HK, Johansson T, Nino AJ, See K, Krohn K, Garcia-Hernandez PA, Recknor CP, Einhorn TA, Dalsky GP, Mitlak BH, Fierlinger A, Lakshmanan MC. Teriparatide for acceleration of fracture repair in humans: a prospective, randomized, double-blind study of 102 postmenopausal women with distal radial fractures. J Bone Miner Res. 2010 Feb;25(2):404-14. doi: 10.1359/jbmr.090731. PMID 19594305
- [Background] Miller PD, Hattersley G, Riis BJ, Williams GC, Lau E, Russo LA, Alexandersen P, Zerbini CA, Hu MY, Harris AG, Fitzpatrick LA, Cosman F, Christiansen C; ACTIVE Study Investigators. Effect of Abaloparatide vs Placebo on New Vertebral Fractures in Postmenopausal Women With Osteoporosis: A Randomized Clinical Trial. JAMA. 2016 Aug 16;316(7):722-33. doi: 10.1001/jama.2016.11136. PMID 27533157
- [Background] Bernhardsson M, Aspenberg P. Abaloparatide versus teriparatide: a head to head comparison of effects on fracture healing in mouse models. Acta Orthop. 2018 Dec;89(6):674-677. doi: 10.1080/17453674.2018.1523771. Epub 2018 Oct 18. PMID 30334479
- [Background] Lanske B, Chandler H, Pierce A, Brown J, Ominsky M, Kostenuik P, Hattersley G. Abaloparatide, a PTH receptor agonist with homology to PTHrP, enhances callus bridging and biomechanical properties in rats with femoral fracture. J Orthop Res. 2019 Apr;37(4):812-820. doi: 10.1002/jor.24254. Epub 2019 Mar 21. PMID 30790359